CLINICAL TRIAL: NCT04349488
Title: Transcranial Direct Current Stimulation Improves Walking and Balance in Acute Stroke Patients - a Randomized, Double-blind, Sham-controlled Study
Brief Title: Transcranial Direct Current Stimulation Acute Stroke Walking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/287
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Acute Stroke
Keywords: Acute Stroke; tDCS; Anodal; Balance; Walking
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: One group receives anodal tDCS, one placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Anode placed over the affected primary motor cortex, cathode over contralateral supra orbital area. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Anodal Transcranial Direct Current Stimulation
- Placebo (Placebo Comparator): Anode montage but current is ramped up over 15 secondes, then ramped down. 2 mA, 20min stimulation, 5 days a week for 4 weeks
  Interventions: Device: Anodal Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Anodal Transcranial Direct Current Stimulation — Subjects received a micro-current through their scalp to induce cortical and subcortical changes
  Other Names: tDCS

SUMMARY:
16 acute stroke patients will be split into 2 groups. One group will receive the real treatment (anodal tDCS) and one group sham.

Subjects will receive, in addition to conventional rehabilitation, 2mA for 20 mins of their attributed tDCS, 5 times a week.

Evaluations will take place before the first stimulation period (48h post stroke), after 1, 2, 3 and 4 weeks.

The evaluations are the Four Square Step Test, the Berg Balance Scale, the Postural Assessment Scale For Stroke, the Trunk Impairment Scale, the Time Up & Go and the 10 meter walking test.

ELIGIBILITY:
Inclusion Criteria:

* First Ever Stroke
* Motor or sensory deficit
* Understands and follows orders
* Signed inform consent

Exclusion Criteria:

• One Yes on the medium and high risk sections of the TSST (Bornheim et al.,2019)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes Four Square Step Test | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  The subject is required to sequentially step over four canes set-up in a cross configuration on the ground. The faster the score, the better the patients balance and coordination.
Changes Berg Balance Scale | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  Balance Test. Minimum score is 0, maximum 36. The higher the score, the better the balance.
Changes Postural Assessment Scale For Stroke | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  alance Test. Minimum score is 0, maximum 56. The higher the score, the better the balance.
Changes Trunk Impairment Scale | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  alance Test. Minimum score is 0, maximum 23. The higher the score, the better the balance.
Changes Time Up & Go | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  To determine fall risk and measure the progress of balance, sit to stand and walking. The faster, the better.
Changes 10 meter walking test | Pre Stimulation (48 hours post stroke), Week 1, Week 2, Week 3, Week 4
  10 meter walking test, the faster the better

CONTACTS AND LOCATIONS:
Locations (1):
- Liege Univeristy Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bornheim S, Croisier JL, Maquet P, Kaux JF. Proposal of a New Transcranial Direct Current Stimulation Safety Screening Tool. Am J Phys Med Rehabil. 2019 Jul;98(7):e77-e78. doi: 10.1097/PHM.0000000000001096. No abstract available. PMID 30431445